CLINICAL TRIAL: NCT03925376
Title: Prognostic Factors of Patients Undergoing Redo Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PURSUE
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Redo Cardiac Surgery
Keywords: Redo cardiac surgery; Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Redo cardiac surgery — Redo cardiac surgery is technically challenging due to scarring of tissues resulting in loss of tissue planes, adhesions, multiple comorbid factors and risk of injury during re-entry.Suggested techniques in coronary artery surgery with a left internal mammary artery include routing the graft through a slit in the pericardium to minimize the possibility of adherence to the sternal table.

SUMMARY:
This study aims to investigate the prognostic significance of baseline characteristics for patients undergoing redo cardiac surgery.

DETAILED DESCRIPTION:
Redo cardiac surgery is associated with an increased risk of postoperative morbidity and mortality. Patients undergoing redo cardiac surgery are becoming increasingly complex due to multiple comorbidities, adherence of mediastinal structures to the undersurface of the sternum as well as the spatial location of patent bypass grafts relative to the route of entry. Association estimates between baseline characteristics and outcomes in those cohort are imprecise. The aim of this study is to identify prognostic factors associated with redo cardiac surgery which may help physicians predict clinical outcomes and guide their treatment decision.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing redo cardiac surgery

Exclusion Criteria:

* Age <18 years;
* Patients with a DNR order or "do not escalate care" order.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Redo cardiac surgery is associated with an increased risk of postoperative morbidity and mortality. Patients undergoing redo cardiac surgery are becoming increasingly complex due to multiple comorbidities, adherence of mediastinal structures to the undersurface of the sternum as well as the spatial location of patent bypass grafts relative to the route of entry.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-04-21 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  Death from any cause at 28 days

SECONDARY OUTCOMES:
60- and 90-day mortality | 60 days and 90 days
  Death from any cause at 60- and 90-days

OTHER OUTCOMES:
Length of stay in the ICU | up to 90 days
  the length of stay in the ICU
Length of stay in the hospital | up to 90 days
  the length of stay in the hospital
Percentage of participants with adverse events | up to 90 days
  Adverse events includes haemorrhage; need for intraoperative/postoperative intra-aortic balloon pumping (IABP); prolonged intubation; acute kidney injury or need for continuous renal replacement therapy (CRRT); poor neurological outcome; infection events

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital, Fudan university, Shanghai, China